CLINICAL TRIAL: NCT07268326
Title: PLATE: Health Effects of Plant-Based Diet in Patients With Rheumatoid Arthritis
Brief Title: Plant-Based Diet for Patients With Rheumatoid Arthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Clinical Research and Prevention (Network)
Collaborators: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Allan Linneberg, Professor, MD, Center for Clinical Research and Prevention
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: H-25045516
Record Dates: First submitted 2025-11-18; First posted 2025-12-05 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: Rheumatoid Arthritis; Plant-based; Dietary intervention; Clinical nutrition
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Diet, Plant-Based

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Care Provider
Masking Description: Project nurses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Other: Plant-based diet
- Control group (No Intervention)

INTERVENTIONS:
Other: Plant-based diet — The intervention is a 100% plant-based diet, and a daily multivitamin supplement. Participants in the intervention group will receive weekly food delivery to their household. Moreover, they will participate in a practical cooking workshop with other participants of the intervention group. Furthermore, they will have three online supervisions with relevant project staff.
  Arms: Intervention group

SUMMARY:
The goal of this clinical trial is to evaluate the effect of a plant-based diet (PBD) intervention in adults with Rheumatoid Arthritis (RA) on disease activity.

The investigators hypothesize that if patients with RA follow a 100% PBD over a 16-week period it will lead to improvements in:

- Disease activity (measured by DAS28), including reduction in symptoms and overall improvements in health-related quality of life.

The effects of the PBD will be compared to a habitual diet, that includes no dietary changes.

Participants in the intervention group will:

* Receive weekly delivery of food boxes which include plant-based food items
* Receive a daily multivitamin supplement
* Receive continuous dietetic guidance
* Participate in a practical cooking class to get an introduction to a PBD
* Participate in three online supervisions throughout the intervention period

Participants in the control group will follow the same plan for the project visits at the hospital but will be restricted to continue their habitual diet. Thus, not performing any dietary changes.

DETAILED DESCRIPTION:
Rheumatoid Arthritis (RA) is a chronic, autoimmune disease, requiring lifelong medical treatment. Evidence has suggested that supporting patients with RA to take an active role in their management of their disease can improve the patients' overall health and quality of life. In addition, patients often ask for support to identify effective ways to reduce symptoms, which include lifestyle changes, of which nutrition may be important. From a patient perspective, the lack of consistent evidence on nutrition also affects patients' choices regarding diet. Patients with RA have expressed that their is insufficient guiding regarding dietary choices. Hypotheses about the effect of various diets on disease activity in RA have been suggested, hence, the influence of pro-inflammatory and anti-inflammatory ingredients have been clinically investigated, however, with very limited studies investigating the effect of a 100% plant-based diet (PBD) on disease activity in RA.

The objective of this study is to investigate if 16-weeks of PBD reduces disease activity and RA-related symptoms, and improves cardio-metabolic health, physical function, mental health, sleep quality and health-related quality of life (HRQoL) in patients with RA.

Thus, in this RCT the patients in the intervention group will be instructed to adhere to a 100% PBD and without changing e.g., exercise habits.

The 16-week intervention consists of

* Weekly delivery of food boxes including plant-based food items for the entire household. Including various different recipes for a balanced PBD.
* A daily multivitamin supplement.
* Continuous dietetic guidance either in person, by phone or e-mail.
* The patients will participate in a practical cooking class to get an introduction to a PBD. Here they will be in groups of approx. 5-8 patients.
* Throughout the intervention period the patients will in addition participate in three online supervisions with the same group they were together with in the cooking class.
* The patients will register their food and drink intake two days before each project visit.

The control group will be asked to maintain habitual diet. At study end, they will receive the same recipes as the intervention group.

All participants, despite group allocation will undergo the same outcome assessments at each project visits (baseline, week 6, week 12, week 16 (end of intervention), and a follow-up visit 12 months after end of intervention:

The following data will be collected:

Baseline:

* Assessment of swollen and tender joints
* Ultrasound of joints
* Patient-reported outcomes (questionnaires)
* Blood samples
* Urine samples
* Feces samples
* Blood pressure
* Anthropometrics (body composition)
* Dietary records

Week 6 and 12:

* Blood samples
* Urine samples
* Dietary records

Week 16:

* Assessment of swollen and tender joints
* Ultrasound of joints
* Patient-reported outcomes (questionnaires)
* Blood samples
* Urine samples
* Feces samples
* Blood pressure
* Anthropometrics (body composition)
* Dietary records

  1-year follow-up:
* Assessment of swollen and tender joints
* Ultrasound of joints
* Patient-reported outcomes (questionnaires)
* Blood samples
* Urine samples
* Feces samples
* Blood pressure
* Anthropometrics (body composition)
* Dietary records

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* DAS28 score ≤3.2, and without swollen joints
* RA diagnosis of minimum one year
* Stable pharmacological treatment for at least four months and with no planned change in treatment within eight weeks

Exclusion Criteria:

* Smokers
* Diabetes mellitus
* Pregnancy / planned pregnancy
* Prednisolone treatment
* DAS28 above 3.2
* Current dietary habits resembling intervention diet (e.g., PBD lifestyle)
* Food allergies and intolerances
* Unable to understand the informed consent and study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Disease activity measured by DAS28 | 16 weeks
  The Disease Activity Score 28 (DAS28) is a composite index used to assess disease activity in patients with rheumatoid arthritis. The DAS28 is a quantification of tender and swollen joints within the hands, shoulders, elbows, wrists, and knees. These assessments, in conjunction with CRP values obtained from blood samples and the self-reported global Visual Analog Scale (VAS) score, will be incorporated into the computation of DAS28. The DAS28 ranges from 0 to 10, with higher scores indicating higher disease activity.

SECONDARY OUTCOMES:
Ultrasound - supportive of the primary outcome | 16 weeks
  Ultrasound is performed bilaterally of the radio-carpal, inter-carpal and radio-ulna joint (with the highest of the 3 scores as the final score for the wrist joint), 1-5 metacarpophalangeal joint (MCP), 2-5 proximal interphalangeal joint (PIP), interphalangeal joint, ankle joint and 2-5 metatarsophalangeal joint (MTP).

OTHER OUTCOMES:
Inflammatory biomarkers | 16 weeks
  Measured in blood samples, including: C-reactive protein (CRP), IL-6 and Soluble urokinase plasminogen activator receptor (suPAR).
Cholesterol | 16 weeks
  Measured by blood samples: Total cholesterol, High-density lipoprotein , Low-density lipoprotein, Very-low density lipoprotein.
Glucose | 16 weeks
  Blood samples of HbA1C
Blood pressure | 16 weeks
  Blood pressure (systolic and diastolic) will be measured, after 5 to 10 minutes of rest with the participant in a sitting/lying position. The blood pressure will be measured three times at the right upper arm, and the average of the three measurements will be documented.
Height | 16 weeks
  Height measured in cm to calculate BMI that will be reported in in kg/m^2
Body composition measured by TANITA weight | 16 weeks
  Participants are weight using TANITA body composition analyzer BC-420MA. The scale also calculates fat%, fat mass (kg), fat free mass (kg), and muscle mass (kg), all details will be obtained.
Waist- and hip circumference | 16 weeks
  Weight, waist- and hip circumference measured in cm to document the ratio
Physical function | 16 weeks
  The Multidimensional Health Assessment Questionnaire (MD-HAQ) is applied to measure self-reported functional status over the previous seven days on ten questions covering dressing, rising, eating, walking, hygiene, reach, grip and everyday activities. The reporting of the results from this questionnaire will cover all these markers that ends up in one total combined score. This is in accordance with the validated questionnaire on how to report the combined result.
  Ref. Pincus, T., Swearingen, C., & Wolfe, F. (1999). Toward a multidimensional Health Assessment Questionnaire (MDHAQ): assessment of advanced activities of daily living and psychological status in the patient-friendly health assessment questionnaire format. Arthritis & Rheumatism: Official Journal of the American College of Rheumatology, 42(10), 2220-2230.
Health-related quality of life (HRQoL) | 16 weeks
  The EuroQuality of Life (EQ-5D) generic health index will be used as a health index to calculate the health-related quality of life.
  The questionnaire comprises a five-part questionnaire. The total sum of these questionnaire will be reported in a total score.
  Ref. Ramos-Goni, Juan M., et al. Quality control process for EQ-5D-5L valuation studies. Value in health, 2017, 20.3: 466-473.
Health-related quality of life by the visual analogue self-rating scale | 16 weeks
  The EuroQuality of Life (EQ-5D) generic health index include a visual analogue self-rating scale. The visual analogue self-rating scale ranges from 0-100. 0 being the worst case scenario, and 100 being best case scenario.
  Ref. Ramos-Goni, Juan M., et al. Quality control process for EQ-5D-5L valuation studies. Value in health, 2017, 20.3: 466-473.
Fatigue | 16 weeks
  Bristol Rheumatoid Arthritis Fatigue (BRAF MDQ). The BRAF MDQ covers several questions of fatigue, including living, cognitive, emotional and physical fatigue. 20 questions are included in the questionnaire, where the total fatigue score will be reported.
  Ref. Primdahl J, Esbensen BA, Pedersen AK, Bech B, de Thurah A. Validation of the Danish versions of the Bristol Rheumatoid Arthritis Fatigue Multi-Dimensional Questionnaires (BRAFs). Scandinavian Journal of Rheumatology. 2021;50(5):351-9.
Pain by Visual Analogue Scale | 16 weeks
  Participants' pain levels will be measured by the Visual Analogue Scale (VAS), which transforms the subjective experience of pain to a measurable quantity. The scale ranges from 0-100. A score of 0 corresponds to the best case scenario of no pain, whereas a score of 100 is the worst possible pain. The result will be reported as a nummeric value.
  Ref: Price DD, McGrath PA, Rafii A, Buckingham B. The validation of visual analogue scales as ratio scale measures for chronic and experimental pain. Pain. 1983;17(1):45-56.
Sleep quality | 16 weeks
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire that assesses sleep quality and disturbances using 24 different questions.
  The reporting of the results from this questionnaire will cover all these questions that ends up in one total combined score. This is in accordance with the validated questionnaire on how to report the combined result.
  Ref. Nicassio PM, et al. Confirmatory factor analysis of the Pittsburgh Sleep Quality Index in rheumatoid arthritis patients. Behav Sleep Med. 2014;12(1):1-12.
Mental health | 16 weeks
  The Hospital Anxiety and Depression Scale (HADS) is used to screen for psychological distress in medical outpatients through self-report. It is a 14-item self-report questionnaire that measures the presence of symptoms related to both anxiety and depression during the past week.
  The reporting of the results from this questionnaire will cover all these questions that ends up in one total combined score. This is in accordance with the validated questionnaire on how to report the combined result.
  Ref. Zigmond, Anthony S.; SNAITH, R. Philip. The hospital anxiety and depression scale. Acta psychiatrica scandinavica, 1983, 67.6: 361-370.
Micronutrient status | 16 weeks
  Changes in nutritional status are measured by biomarkers in blood to assess micronutrient status of 25-hydroxy-vitamin D, ionized calcium, B12, vitamin K, zinc, iron, folate.
Electrolyte status | 16 weeks
  Changes in nutritional status are measured by electrolytes in the blood of natrium and potassium.
Dietary intake measured by spot urine | 16 weeks
  Changes in dietary status are measured by biomarkers in spot urine, including urea, creatinine, nitrogen, potassium, natrium, and pH, hippuric acid, hydroxyhippuric acid, dihydrocaffeic acid sulfate.
Gut microbiome | 16 weeks
  Changes in gut microbiome are measured in feces, by looking at the gut microbiome composition, short chain fatty acids, and bile salt.

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Bispebjerg and Frederiksberg Hospital, Center for Clinical Research and Prevention, Frederiksberg
  - The Department of Rheumatology and Spine Diseases, Copenhagen Center for Arthritis Research (COPECARE), Rigshospitalet, Glostrup, Glostrup Municipality

IPD SHARING:
Plan to Share IPD: No